CLINICAL TRIAL: NCT03238911
Title: A Randomized, Open-label, Comparative Trial Comparing the Incidence of Hypophosphatemia in Relation to Treatment With Iron Isomaltoside/Ferric Derisomaltose and Ferric Carboxymaltose in Subjects With Iron Deficiency Anaemia (Phosphare-IDA-04)
Brief Title: Incidence of Hypophosphatemia After Treatment With Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose in Subjects With Iron Deficiency Anaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IDA-04
Record Dates: First submitted 2017-07-06; First posted 2017-08-03 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Iron Deficiency Anaemia; Iron Deficiency Anemia
Keywords: Iron Deficiency Anaemia; Iron Deficiency Anemia; IDA; Intravenous iron replacement therapy; Iron deficiency; Iron isomaltoside; Ferric derisomaltose; Monofer; Monoferric; Monover; Monofar; Monoferro; Hypophosphatemia; Ferric carboxymaltose
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies; Hypophosphatemia | interventions — iron isomaltoside 1000; ferric derisomaltose; ferric carboxymaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iron isomaltoside/ferric derisomaltose (Experimental): Administered IV
  Interventions: Drug: Iron isomaltoside/ferric derisomaltose
- Ferric carboxymaltose (Active Comparator): Administered IV
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Iron isomaltoside/ferric derisomaltose — Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  The dose of iron isomaltoside/ferric derisomaltose for the individual subject was a single IV infusion of 1000 mg (10 mL containing 1000 mg iron isomaltoside/ferric derisomaltose diluted in 100 mL 0.9 % sodium chloride), given over approximately 20 minutes (50 mg iron/min) at baseline (cumulative dose: 1000 mg).
  Other Names: Monofer®, Monoferric®, Monover®, Monofar®, Monoferro®
  Arms: Iron isomaltoside/ferric derisomaltose
Drug: Ferric carboxymaltose — Ferric carboxymaltose (Injectafer®; 50 mg/mL) was the comparator in this trial.
  Ferric carboxymaltose was administered as 750 mg, infused over at least 15 minutes at baseline and on day 7 (cumulative dose: 1500 mg).
  Other Names: Injectafer®, Ferinject®
  Arms: Ferric carboxymaltose

SUMMARY:
The trial was designed to evaluate the incidence of unintended hypophosphatemia (low level of phosphate in the blood) in subjects with iron deficiency anaemia (IDA).

DETAILED DESCRIPTION:
This trial was designed to evaluate the effect of IV iron isomaltoside/ferric derisomaltose compared with IV ferric carboxymaltose on s-phosphate in subjects with IDA caused by different etiologies.

The subjects received either a single intravenous (IV) dose of iron isomaltoside/ferric derisomaltose (1000 mg at baseline) or two IV doses of ferric carboxymaltose (one dose 750 mg at baseline and a second dose 750 mg on day 7; cumulative dose: 1500 mg). The study subjects were monitored for up to 35 days from baseline.

ELIGIBILITY:
Inclusion Criteria include:

* Subjects diagnosed with IDA, caused by different aetiologies
* Haemoglobin (Hb) ≤ 11 g/dL
* Body weight > 50 kg
* Serum ferritin (S-ferritin) < 100 ng/mL
* Estimated glomerular filtration rate (eGFR) ≥ 65 mL/min/1.73 m2
* Serum phosphate (S-phosphate) > 2.5 mg/dL
* Intolerance or unresponsiveness to oral iron
* Willingness to participate and signing the Informed Consent Form (ICF)

Exclusion Criteria include:

* Acute bleeding > 500 mL within 72 hours
* Anaemia predominantly caused by factors other than IDA
* Hemochromatosis or other iron storage disorders
* Previous serious hypersensitivity reactions to any IV iron compounds
* Treatment with IV iron within the last 30 days prior to screening
* Treatment with erythropoietin or erythropoietin-stimulation agents
* Red blood cell transfusion, radiotherapy, and/or chemotherapy
* Received an investigational drug within the last 30 days prior to screening
* Planned surgical procedure within the trial period
* Hepatic enzymes > 3 times upper limit of normal
* Surgery under anaesthetic within the last 30 days prior to screening
* Any non-viral infection within the last 30 days prior to screening
* Alcohol or drug abuse within the past 6 months
* Vitamin D deficiency
* Untreated hyperparathyroidism
* Kidney transplantation
* Active malignant disease, disease-free for less than 5 years
* History of a psychological illness or seizures
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 123 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S Clinical and Non-clinical Research, Study Director — Pharmacosmos A/S
Locations (14):
- United States (14):
  - Pharmacosmos Investigational Site, Los Angeles, California
  - Pharmacosmos Investigational Site, Sacramento, California
  - Pharmacosmos Investigational Site, Santa Ana, California
  - Pharmacosmos Investigational Site, Clearwater, Florida
  - Pharmacosmos Investigational Site, Miami, Florida
  - Pharmacosmos Investigational Site 1, Miami, Florida
  - Pharmacosmos Investigational Site 2, Miami, Florida
  - Pharmacosmos Investigational Site, Indianapolis, Indiana
  - Pharmacosmos Investigational Site, Wichita, Kansas
  - Pharmacosmos Investigational Site, Metairie, Louisiana
  - Pharmacosmos Investigational Site, Lancaster, Pennsylvania
  - Pharmacosmos Investigational Site, Houston, Texas
  - Pharmacosmos Investigational Site, Orem, Utah
  - Pharmacosmos Investigational Site, Leesburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wolf M, Rubin J, Achebe M, Econs M, Peacock M, Imel E, Thomsen L, Carpenter T, Weber T, Zoller H. Effects of iron isomaltoside versus ferric carboxymaltose on hormonal control of phosphate homeostasis: The PHOSPHARE-IDA04/05 randomized controlled trials. Journal of the Endocrine Society, Volume 3, Issue Supplement_1, April-May 2019, OR13-3, https://doi.org/10.1210/js.2019-OR13-3
- [Derived] Wolf M, Rubin J, Achebe M, Econs MJ, Peacock M, Imel EA, Thomsen LL, Carpenter TO, Weber T, Brandenburg V, Zoller H. Effects of Iron Isomaltoside vs Ferric Carboxymaltose on Hypophosphatemia in Iron-Deficiency Anemia: Two Randomized Clinical Trials. JAMA. 2020 Feb 4;323(5):432-443. doi: 10.1001/jama.2019.22450. PMID 32016310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 310 subjects were screened and 123 subjects were randomised into the trial.
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  Subjects received iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) as a single IV infusion of 1000 mg at the baseline visit.
- Ferric Carboxymaltose: Ferric carboxymaltose (Injectafer®; 50 mg/mL) was the comparator product in this trial.
  The dose of ferric carboxymaltose for the individual subject was 750 mg, infused IV at baseline and on day 7 (cumulative dose: 1500 mg).
Period: Overall Study
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Started | 62 | 61
Safety Analysis Set | 63 (1 subject from ferric carboxymaltose group received iron isomaltoside/ferric derisomaltose in error.) | 60 (1 subject from ferric carboxymaltose group received iron isomaltoside/ferric derisomaltose in error.)
Completed | 59 | 58
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose, administered IV
- Ferric Carboxymaltose: Ferric carboxymaltose, administered IV
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose | Total
Number analyzed (Participants) | 63 | 60 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 54 | 114
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.4) | 46.3 (11.6) | 45.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 57 | 118
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 36 | 73
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 19 | 41
  White | 38 | 38 | 76
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/American Indian | 0 | 1 | 1
  White/American Indian | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 63 | 60 | 123
Iron Deficiency Anaemia (IDA) due to gynaecological blood loss [Count of Participants; unit: Participants]
  Yes | 41 | 42 | 83
  No | 22 | 18 | 40
Current smoker [Count of Participants; unit: Participants]
  Yes | 6 | 8 | 14
  No | 57 | 52 | 109
S-phosphate level at screening [Count of Participants; unit: Participants]
  <3.5 mg/dL | 32 | 33 | 65
  ≥3.5 mg/dL | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypophosphatemia (S-phosphate Level <2 mg/dL)
Description: Safety
  The incidence of hypophosphatemia (defined as s-phosphate <2 mg/dL) at any time from baseline up to day 35.
Time Frame: Baseline to day 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
Participants | 5 | 45
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Power: The power was set to 80%. Assuming incidences of 15% for iron isomaltoside/ferric derisomaltose and 40% for ferric carboxymaltose, 49 subjects in each treatment group were required to detect a difference between the treatment groups. The significance level was set to 5%; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = -67.0, 95% CI 2-sided [-77.4 to -51.5] — Iron isomaltoside/ferric derisomaltose was compared to ferric carboxymaltose by estimation of the risk difference and the associated 95% CI, adjusting for strata (underlying disease and screening s-phosphate) using the Cochran-Mantel-Haenszel method

2. Secondary Outcome: Time With Hypophosphatemia ( S-phosphate Level <2.0 mg/dL)
Description: Safety
  Time with hypophosphatemia (i.e. time with s-phosphate level < 2.0 mg/dL) from baseline up to day 35.
  The time with hypophosphatemia was calculated as the actual number of days from the first day where s-phosphate was <2 mg/dL until the first day when s-phosphate was ≥2 mg/dL. If the subject did not reach s-phosphate ≥2 mg/dL, the subject was regarded as censored on day 35.
Time Frame: Baseline to day 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
days | 15 [7 to 56] | 29 [21 to 42]
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; The time with hypophosphatemia from baseline to day 35 was estimated by a Kaplan-Meier plot. The treatment groups were compared by a log-rank test. Only subjects who had one or more s-phosphate value(s) <2 mg/dL were included; Test type: Superiority; p = 0.8979, Log Rank

3. Secondary Outcome: Proportion of Subjects With Hypophosphatemia on Day 35 ( S-phosphate Level <2.0 mg/dL)
Description: Safety
  Evaluate the proportion of subjects with hypophosphatemia (s-phosphate level <2.0 mg/dL) on day 35.
Time Frame: Baseline to day 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 59 | 58
Participants | 1 | 24
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Iron isomaltoside/ferric derisomaltose will be compared to ferric carboxymaltose by estimation of the risk difference and the associated 95 % CI, adjusting for strata (type of underlying disease (women with IDA due to gynaecological blood losses; yes/no) and screening s-phosphate level (< or ≥ 3.5 mg/dL)) using the Cochran-Mantel-Haenszel method; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Risk Difference (RD) = -39.2, 95% CI 2-sided [-52.2 to -23.3]

4. Secondary Outcome: Absolute [∆] Changes in S-phosphate From Baseline to Day 1, 7, 8, 14, 21, and 35
Description: Safety
  Absolute [∆] changes in s-phosphate from baseline to day 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
mg/dL
  Day 1: number analyzed (Participants) | 59 | 57
  Day 1 | 0.25 (0.55) | -0.24 (0.61)
  Day 7: number analyzed (Participants) | 60 | 58
  Day 7 | -0.06 (0.75) | -1.15 (0.63)
  Day 8: number analyzed (Participants) | 57 | 57
  Day 8 | -0.10 (0.77) | -1.15 (0.64)
  Day 14: number analyzed (Participants) | 58 | 56
  Day 14 | -0.04 (0.75) | -1.44 (0.83)
  Day 21: number analyzed (Participants) | 54 | 56
  Day 21 | 0.04 (0.69) | -1.02 (0.99)
  Day 35: number analyzed (Participants) | 59 | 58
  Day 35 | 0.24 (0.76) | -0.92 (0.85)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 1 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.31 to 0.65]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 7 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [0.85 to 1.27]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 8 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.81 to 1.25]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 14 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [1.10 to 1.60]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 21 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 1.03, 95% CI 2-sided [0.75 to 1.32]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; Day 35 Change from baseline was analysed using a Restricted Maximum Likelihood (REML)-based Mixed Model for Repeated Measures (MMRM) approach. All subjects with post-baseline data were included with their observed data. The model included the fixed, categorical effects of treatment, strata, day, treatment-by-day interaction, as well as the continuous, fixed covariates of the parameters baseline value, and baseline value-by-day interaction; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 1.13, 95% CI 2-sided [0.86 to 1.39]

5. Secondary Outcome: Relative [%] Changes in S-phosphate From Baseline to Day 1, 7, 8, 14, 21, and 35
Description: Safety
  Relative [%] changes in s-phosphate from baseline to day 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
Percentage change from baseline
  Day 1: number analyzed (Participants) | 59 | 56
  Day 1 | 9.31 (18.98) | -5.94 (16.59)
  Day 7: number analyzed (Participants) | 60 | 58
  Day 7 | 0.55 (23.15) | -33.68 (17.53)
  Day 8: number analyzed (Participants) | 57 | 57
  Day 8 | -0.95 (24.02) | -34.03 (17.61)
  Day 14: number analyzed (Participants) | 58 | 56
  Day 14 | 1.13 (25.21) | -42.59 (24.81)
  Day 21: number analyzed (Participants) | 54 | 56
  Day 21 | 2.85 (22.66) | -30.11 (30.79)
  Day 35: number analyzed (Participants) | 59 | 58
  Day 35 | 9.69 (24.55) | -27.58 (27.47)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 15.55, 95% CI 2-sided [10.32 to 20.79]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 33.23, 95% CI 2-sided [26.62 to 39.84]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 32.78, 95% CI 2-sided [25.71 to 39.84]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 42.11, 95% CI 2-sided [33.89 to 50.32]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 32.28, 95% CI 2-sided [23.09 to 41.48]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 36.06, 95% CI 2-sided [27.33 to 44.78]

6. Secondary Outcome: Change From Baseline in Fractional Phosphate Urinary Excretion
Description: Safety
  Change in absolute fractional phosphate urinary excretion from baseline to days 1, 7, 8, 14, 21, and 35.
  Fractional excretion of phosphate (FEPi) is calculated as ([phosphate in urine X creatinine in serum]/[phosphate in serum X creatinine in urine]) X 100, and the unit is %.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: percentage excreted
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
percentage excreted
  Day 1: number analyzed (Participants) | 36 | 38
  Day 1 | -1.73 (4.85) | 2.44 (5.09)
  Day 7: number analyzed (Participants) | 38 | 40
  Day 7 | 0.56 (8.30) | 8.12 (9.16)
  Day 8: number analyzed (Participants) | 35 | 40
  Day 8 | 1.21 (7.71) | 9.08 (11.30)
  Day 14: number analyzed (Participants) | 35 | 40
  Day 14 | 0.10 (7.34) | 11.46 (13.53)
  Day 21: number analyzed (Participants) | 32 | 40
  Day 21 | 0.78 (9.46) | 9.43 (12.33)
  Day 35: number analyzed (Participants) | 36 | 41
  Day 35 | -1.97 (7.29) | 4.90 (11.07)

7. Secondary Outcome: Change in Concentration of (Intact) Fibroblast Growth Factor 23 (iFGF23) From Baseline to Day 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in concentration of (Intact) Fibroblast Growth Factor 23 (iFGF23) from baseline to day 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
pg/mL
  Day 1: number analyzed (Participants) | 55 | 56
  Day 1 | -2.7 (28.6) | 103.6 (89.5)
  Day 7: number analyzed (Participants) | 56 | 54
  Day 7 | 6.8 (26.9) | 70.3 (78.4)
  Day 8: number analyzed (Participants) | 50 | 54
  Day 8 | 4.9 (25.2) | 305.9 (262.3)
  Day 14: number analyzed (Participants) | 53 | 54
  Day 14 | -8.6 (25.7) | 106.1 (114.9)
  Day 21: number analyzed (Participants) | 50 | 53
  Day 21 | -0.9 (39.7) | 66.7 (96.6)
  Day 35: number analyzed (Participants) | 54 | 55
  Day 35 | -10.5 (25.6) | 34.7 (64.2)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -105.74, 95% CI 2-sided [-131.04 to -80.45]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -60.76, 95% CI 2-sided [-82.95 to -38.58]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -293.23, 95% CI 2-sided [-368.15 to -218.30]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -117.47, 95% CI 2-sided [-151.60 to -83.33]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -71.21, 95% CI 2-sided [-101.80 to -40.61]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -37.16, 95% CI 2-sided [-54.92 to -19.39]

8. Secondary Outcome: Change in C-terminal Fibroblast Growth Factor 23 (cFGF23) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in C-terminal Fibroblast Growth Factor 23 (cFGF23) from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: RU/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
RU/mL
  Day 1: number analyzed (Participants) | 56 | 52
  Day 1 | -742.3 (800.7) | -390.2 (665.7)
  Day 7: number analyzed (Participants) | 53 | 51
  Day 7 | -723.6 (801.6) | -477.5 (652.0)
  Day 8: number analyzed (Participants) | 52 | 51
  Day 8 | -648.9 (757.5) | -284.2 (638.6)
  Day 14: number analyzed (Participants) | 54 | 51
  Day 14 | -717.9 (798.2) | -401.5 (661.5)
  Day 21: number analyzed (Participants) | 48 | 49
  Day 21 | -678.1 (783.5) | -458.9 (658.9)
  Day 35: number analyzed (Participants) | 50 | 53
  Day 35 | -660.1 (806.7) | -481.3 (653.7)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -99.1, 95% CI 2-sided [-136.42 to -61.76]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -49.3, 95% CI 2-sided [-72.80 to -25.90]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -191.3, 95% CI 2-sided [-242.47 to -140.09]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -100.7, 95% CI 2-sided [-137.19 to -64.20]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -48.4, 95% CI 2-sided [-71.78 to -24.96]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.1411, Mixed model for repeated measures; Mean Difference (Final Values) = -15.0, 95% CI 2-sided [-35.04 to 5.06]

9. Secondary Outcome: Change in Vitamin 25-Hydroxyvitamin D (Vitamin D 25) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in vitamin 25-Hydroxyvitamin D (vitamin D 25) from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
ng/mL
  Day 1: number analyzed (Participants) | 58 | 59
  Day 1 | 0.04 (2.26) | 0.32 (2.26)
  Day 7: number analyzed (Participants) | 59 | 57
  Day 7 | 0.81 (3.34) | -0.94 (3.93)
  Day 8: number analyzed (Participants) | 57 | 58
  Day 8 | 0.32 (3.35) | -0.07 (5.07)
  Day 14: number analyzed (Participants) | 57 | 57
  Day 14 | 0.71 (5.17) | -1.29 (5.14)
  Day 21: number analyzed (Participants) | 54 | 57
  Day 21 | 0.78 (6.03) | -0.90 (4.70)
  Day 35: number analyzed (Participants) | 58 | 56
  Day 35 | -0.24 (6.44) | -0.72 (4.34)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.5620, Mixed model for repeated measures; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.08 to 0.59]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0126, Mixed model for repeated measures; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [0.38 to 3.12]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.6080, Mixed model for repeated measures; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-1.19 to 2.02]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.0379, Mixed model for repeated measures; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [0.12 to 4.05]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.2368, Mixed model for repeated measures; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [-0.78 to 3.12]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.8287, Mixed model for repeated measures; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-2.18 to 1.75]

10. Secondary Outcome: Change in 1,25-Dihydroxyvitamin D (Vitamin D 1.25) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in 1,25-Dihydroxyvitamin D (vitamin D 1.25) from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
pg/mL
  Day 1: number analyzed (Participants) | 58 | 59
  Day 1 | 5.13 (13.05) | -20.57 (17.56)
  Day 7: number analyzed (Participants) | 59 | 58
  Day 7 | -19.92 (24.57) | -38.84 (20.86)
  Day 8: number analyzed (Participants) | 57 | 58
  Day 8 | -16.07 (25.10) | -39.63 (27.11)
  Day 14: number analyzed (Participants) | 57 | 57
  Day 14 | -3.31 (15.93) | -39.04 (27.46)
  Day 21: number analyzed (Participants) | 55 | 56
  Day 21 | -3.37 (16.45) | -28.89 (30.06)
  Day 35: number analyzed (Participants) | 58 | 58
  Day 35 | -3.86 (20.08) | -17.94 (26.15)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 24.27, 95% CI 2-sided [18.81 to 29.73]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 15.75, 95% CI 2-sided [8.83 to 22.67]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 20.14, 95% CI 2-sided [12.07 to 28.22]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 32.22, 95% CI 2-sided [25.49 to 38.96]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 22.87, 95% CI 2-sided [14.79 to 30.95]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.0043, Mixed model for repeated measures; Mean Difference (Final Values) = 10.60, 95% CI 2-sided [3.39 to 17.82]

11. Secondary Outcome: Change in 24,25-Dihydroxyvitamin D (Vitamin D 24.25) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in 24,25-Dihydroxyvitamin D (vitamin D 24.25) from baseline to days 1, 7, 8, 14, 21, and 35
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
ng/mL
  Day 1: number analyzed (Participants) | 57 | 55
  Day 1 | -0.02 (0.41) | 0.13 (0.51)
  Day 7: number analyzed (Participants) | 58 | 54
  Day 7 | 0.30 (0.49) | 0.72 (0.78)
  Day 8: number analyzed (Participants) | 56 | 54
  Day 8 | 0.19 (0.69) | 0.71 (0.84)
  Day 14: number analyzed (Participants) | 56 | 52
  Day 14 | 0.13 (0.60) | 0.95 (0.98)
  Day 21: number analyzed (Participants) | 54 | 51
  Day 21 | 0.12 (0.93) | 0.75 (0.93)
  Day 35: number analyzed (Participants) | 57 | 54
  Day 35 | 0.06 (0.89) | 0.60 (0.99)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0552, Mixed model for repeated measures; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.34 to 0.00]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0023, Mixed model for repeated measures; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.60 to -0.13]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.0008, Mixed model for repeated measures; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.80 to -0.21]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.11 to -0.49]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0006, Mixed model for repeated measures; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-1.01 to -0.28]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.0014, Mixed model for repeated measures; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.94 to -0.23]

12. Secondary Outcome: Change in Intact Parathyroid Hormone (PTH) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in intact Parathyroid hormone (PTH) from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
pg/mL
  Day 1: number analyzed (Participants) | 57 | 54
  Day 1 | -1.3 (20.2) | 0.7 (21.3)
  Day 7: number analyzed (Participants) | 57 | 56
  Day 7 | -4.6 (26.6) | 7.8 (26.6)
  Day 8: number analyzed (Participants) | 54 | 55
  Day 8 | 1.8 (27.9) | 2.6 (29.2)
  Day 14: number analyzed (Participants) | 55 | 56
  Day 14 | 3.2 (30.6) | 16.7 (33.7)
  Day 21: number analyzed (Participants) | 52 | 55
  Day 21 | -3.1 (22.8) | 17.2 (34.9)
  Day 35: number analyzed (Participants) | 53 | 56
  Day 35 | 0.2 (27.9) | 22.1 (41.2)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.7447, Mixed model for repeated measures; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-7.96 to 5.71]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0363, Mixed model for repeated measures; Mean Difference (Final Values) = -9.70, 95% CI 2-sided [-18.78 to -0.63]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.9242, Mixed model for repeated measures; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-10.56 to 9.59]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.0602, Mixed model for repeated measures; Mean Difference (Final Values) = -11.17, 95% CI 2-sided [-22.84 to 0.49]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0008, Mixed model for repeated measures; Mean Difference (Final Values) = -18.20, 95% CI 2-sided [-28.68 to -7.73]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.0031, Mixed model for repeated measures; Mean Difference (Final Values) = -19.79, 95% CI 2-sided [-32.75 to -6.83]

13. Secondary Outcome: Change in Ionized Calcium From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Safety
  Change in ionized calcium from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
mg/dL
  Day 1: number analyzed (Participants) | 53 | 57
  Day 1 | 0.04 (0.18) | 0.00 (0.20)
  Day 7: number analyzed (Participants) | 52 | 56
  Day 7 | 0.02 (0.16) | -0.07 (0.22)
  Day 8: number analyzed (Participants) | 51 | 56
  Day 8 | 0.03 (0.19) | -0.03 (0.20)
  Day 14: number analyzed (Participants) | 53 | 53
  Day 14 | 0.02 (0.22) | -0.08 (0.22)
  Day 21: number analyzed (Participants) | 50 | 50
  Day 21 | 0.08 (0.19) | -0.03 (0.21)
  Day 35: number analyzed (Participants) | 49 | 55
  Day 35 | 0.02 (0.21) | -0.03 (0.20)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.2670, Mixed model for repeated measures; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.029 to 0.104]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0040, Mixed model for repeated measures; Mean Difference (Final Values) = 0.085, 95% CI 2-sided [0.028 to 0.142]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.0472, Mixed model for repeated measures; Mean Difference (Final Values) = 0.064, 95% CI 2-sided [0.001 to 0.127]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.0050, Mixed model for repeated measures; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.031 to 0.171]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0061, Mixed model for repeated measures; Mean Difference (Final Values) = 0.101, 95% CI 2-sided [0.029 to 0.172]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.1282, Mixed model for repeated measures; Mean Difference (Final Values) = 0.055, 95% CI 2-sided [-0.016 to 0.126]

14. Secondary Outcome: Incidence of Protocol-defined Serious or Severe Hypersensitivity Reactions
Description: Safety
  For this endpoint, the number of participants with serious or severe hypersensitivity reactions were evaluated.
Time Frame: Baseline to day 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 60
Participants | 1 | 0

15. Secondary Outcome: Change in Hemoglobin (Hb) Per Gram Iron From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Efficacy
  Change in hemoglobin (Hb) per gram iron from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Intention-To-Treat (ITT) analysis set: included all randomised subjects.
Measure: Mean (Standard Deviation); unit: g/dL per g of iron
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 62 | 61
g/dL per g of iron
  Day 1: number analyzed (Participants) | 54 | 53
  Day 1 | -0.16 (1.29) | 0.28 (1.82)
  Day 7: number analyzed (Participants) | 54 | 58
  Day 7 | 0.65 (0.86) | 0.94 (1.49)
  Day 8: number analyzed (Participants) | 54 | 55
  Day 8 | 0.50 (1.14) | 0.64 (0.81)
  Day 14: number analyzed (Participants) | 53 | 54
  Day 14 | 1.55 (1.53) | 1.16 (0.90)
  Day 21: number analyzed (Participants) | 53 | 56
  Day 21 | 1.68 (1.40) | 1.44 (0.97)
  Day 35: number analyzed (Participants) | 56 | 56
  Day 35 | 2.16 (1.62) | 1.94 (1.02)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4618, Mixed model for repeated measures; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.82 to 0.37]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.3660, Mixed model for repeated measures; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.54 to 0.20]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.8580, Mixed model for repeated measures; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.25 to 0.30]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.0257, Mixed model for repeated measures; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.05 to 0.74]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0016, Mixed model for repeated measures; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [0.19 to 0.77]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.0185, Mixed model for repeated measures; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.07 to 0.76]

16. Secondary Outcome: Change in S-ferritin From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Efficacy
  Change in s-ferritin from baseline to days 1, 7, 8, 14, 21, and 35.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Intention-To-Treat (ITT) analysis set: included all randomised subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 62 | 61
ng/mL
  Day 1: number analyzed (Participants) | 58 | 59
  Day 1 | 82.0 (58.3) | 94.7 (62.4)
  Day 7: number analyzed (Participants) | 59 | 59
  Day 7 | 261.7 (184.2) | 289.5 (173.0)
  Day 8: number analyzed (Participants) | 57 | 59
  Day 8 | 248.1 (182.4) | 325.8 (220.1)
  Day 14: number analyzed (Participants) | 57 | 57
  Day 14 | 133.9 (109.9) | 352.9 (223.4)
  Day 21: number analyzed (Participants) | 55 | 57
  Day 21 | 97.2 (127.6) | 179.2 (135.0)
  Day 35: number analyzed (Participants) | 58 | 59
  Day 35 | 46.8 (63.0) | 108.9 (107.3)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1922, Mixed model for repeated measures; Mean Difference (Final Values) = -14.84, 95% CI 2-sided [-37.26 to 7.57]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.5601, Mixed model for repeated measures; Mean Difference (Final Values) = -18.28, 95% CI 2-sided [-80.24 to 43.68]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.0459, Mixed model for repeated measures; Mean Difference (Final Values) = -71.02, 95% CI 2-sided [-140.74 to -1.30]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -207.33, 95% CI 2-sided [-268.82 to -145.84]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0010, Mixed model for repeated measures; Mean Difference (Final Values) = -78.60, 95% CI 2-sided [-124.81 to -32.39]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.0002, Mixed model for repeated measures; Mean Difference (Final Values) = -58.79, 95% CI 2-sided [-88.75 to -28.82]

17. Secondary Outcome: Change in Transferrin Saturation (TSAT) From Baseline to Days 1, 7, 8, 14, 21, and 35
Description: Efficacy
  Change in Transferrin Saturation (TSAT) from baseline to days 1, 7, 8, 14, 21, and 35.
  TSAT is the value of serum iron divided by the total iron-binding capacity and the unit is %, which referrers to % of iron-binding sites of transferrin being occupied by iron.
Time Frame: Baseline, days 1, 7, 8, 14, 21, and 35
Population: Intention-To-Treat (ITT) analysis set: included all randomised subjects.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 62 | 61
percentage of saturation
  Day 1: number analyzed (Participants) | 57 | 59
  Day 1 | 118.9 (52.0) | 85.7 (40.4)
  Day 7: number analyzed (Participants) | 58 | 59
  Day 7 | 10.2 (34.8) | 12.9 (11.2)
  Day 8: number analyzed (Participants) | 56 | 59
  Day 8 | 6.3 (34.7) | 61.2 (43.0)
  Day 14: number analyzed (Participants) | 56 | 57
  Day 14 | 4.8 (32.6) | 16.4 (11.3)
  Day 21: number analyzed (Participants) | 54 | 56
  Day 21 | 6.8 (31.1) | 16.6 (11.7)
  Day 35: number analyzed (Participants) | 56 | 59
  Day 35 | 3.1 (32.3) | 14.7 (10.8)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 40.82, 95% CI 2-sided [26.30 to 55.33]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0089, Mixed model for repeated measures; Mean Difference (Final Values) = 6.61, 95% CI 2-sided [1.69 to 11.53]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = -43.48, 95% CI 2-sided [-54.92 to -32.03]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.3730, Mixed model for repeated measures; Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-5.41 to 2.04]
Statistical Analysis 5: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.4778, Mixed model for repeated measures; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-6.15 to 2.90]
Statistical Analysis 6: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; [analysis description as in outcome 4, analysis 6]; Test type: Superiority; p = 0.3575, Mixed model for repeated measures; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-5.44 to 1.98]

18. Post Hoc Outcome: Incidence of S-phosphate Level ≤1.0 mg/dL at Any Time From Baseline to Day 35
Description: Safety
  Incidence of hypophosphatemia (defined as s-phosphate level ≤1 mg/dL) at any time from baseline up to day 35.
Time Frame: Baseline to day 35
Population: Safety analysis set: included all subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
Number analyzed (Participants) | 63 | 59
Participants | 0 | 7
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Ferric Carboxymaltose; The rate difference with 95% Newcombe confidence interval, adjusted for stratum using the Cochran-Mantel-Haenszel method, could not be estimated due to lack of events. Thus, the unadjusted treatment difference is presented together with 95% Wald-based confidence interval. The p-value is based on the Cochran-Mantel-Haenszel statistics; Test type: Superiority; p = 0.0050, Cochran-Mantel-Haenszel; Risk Difference (RD) = -11.9, 95% CI 2-sided [-20.1 to -3.6]

ADVERSE EVENTS:
Time Frame: From the time subjects signed the informed consent form (CRF) and until they completed the study, all adverse events (AEs) or serious adverse events (SAEs) were reported in the CRF. The actual study duration was 35 days (or shorted if the trial was discontinued). Overall, eligible subjects participated in the trial for approximately 9 weeks (including a 28-day screening period).
Description: An AE was described as follows: the nature of the event was described in precise, standard medical terminology (i.e. not necessarily the exact words used by the subject). If known, a specific diagnosis was stated. Furthermore, the Investigator described an AE regarding seriousness, severity, relatedness, and outcome.
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Ferric Carboxymaltose
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/60
Other Adverse Events (participants affected / at risk) | 0/63 | 25/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=63) | Ferric Carboxymaltose (N=60)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=63) | Ferric Carboxymaltose (N=60)
Blood phosphorus decreased (Investigations) | 0 (0) | 13 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 12 (12)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before 1 year after completion of the Study report the Investigator must not publish details regarding the Protocol and the conduct or results of the Trial. However, if a joint publication is submitted for publication the individual Investigator has no right to publish results from his/her centre until such the joint publication is actually issued.

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT03238911/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT03238911/SAP_001.pdf